CLINICAL TRIAL: NCT00871338
Title: Study in Healthy Children of GSK Biologicals' DTPa-IPV/Hib-MenC-TT Vaccine, GSK2197870A, Co-administered With Prevenar™ as a Three-dose Primary Vaccination Course in Infancy Followed by a Booster Dose of Menitorix™ at 12 Months of Age
Brief Title: Study to Evaluate GSK Biologicals' GSK2197870A Vaccine Given as Primary Course in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111709
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-09

CONDITIONS: Neisseria Meningitidis; Haemophilus Influenzae Type b
Keywords: combined; Vaccines
MeSH Terms: conditions — Haemophilus Infections | interventions — Tetanus Toxoid; DTP-IPV-Hib vaccine; Heptavalent Pneumococcal Conjugate Vaccine; diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine

ARMS (2):
- GSK2197870A Group (Experimental): Subjects aged between and including 6 and 12 weeks of age at the time of first vaccination received 3 doses of GSK2197870A vaccine at Months 0, 1 and 2, 2 doses of Prevenar™ vaccine at Months 0 and 2 and a booster dose of Menitorix™ vaccine at Month 10. All vaccines were administered intramuscularly. GSK2197870A and Menitorix™ vaccines were administered in the right upper anterolateral thigh and Prevenar™ vaccine in the left upper anterolateral thigh.
  Interventions: Biological: GSK2197870A; Biological: Prevenar™; Biological: Menitorix™
- Pediacel Group (Active Comparator): Subjects aged between and including 6 and 12 weeks of age at the time of first vaccination received 3 doses of Pediacel™ vaccine at Months 0, 1 and 2, 2 doses of Prevenar™ vaccine at Months 0 and 2, 2 doses of Menjugate™ vaccine at Months 1 and 2 and a booster dose of Menitorix™ at Month 10. All vaccines were administered intramuscularly. Pediacel™ and Menitorix™ vaccines were administered in the right upper anterolateral thigh and Prevenar™ vaccine in the left upper anterolateral thigh and Menjugate™ vaccine in the left lower anterolateral thigh.
  Interventions: Biological: Prevenar™; Biological: Menitorix™; Biological: Pediacel™; Biological: Menjugate™

INTERVENTIONS:
Biological: GSK2197870A — 3 doses given at 2, 3 and 4 months of age
  Other Names: GSK Biologicals' combined diphtheria; tetanus; acellular pertussis; polio; HiB and Neisseria meningitidis serogroup C tetanus toxoid conjugate vaccine.
  Arms: GSK2197870A Group
Biological: Prevenar™ — 3 co-administered doses, intramuscular into right thigh
  Other Names: Pfizer's 13-valent pneumococcal polysaccharide conjugate vaccine
Biological: Menitorix™ — 1 booster dose at 12 months of age
  Other Names: GSK Biologicals' combined Haemophilus influenzae type b and Neisseria meningitidis serogroup C tetanus toxoid conjugate vaccine.
Biological: Pediacel™ — 3 doses given at 2, 3 and 4 months of age
  Other Names: Sanofi-Pasteur-MSD's combined DTPa-inactivated polio-Haemophilus influenzae type b vaccine.
  Arms: Pediacel Group
Biological: Menjugate™ — 2 doses given at 3 and 4 months of age
  Other Names: Novartis' meningococcal serogroup C CRM197 protein conjugated vaccine.
  Arms: Pediacel Group

SUMMARY:
The purpose of this Phase II study is to evaluate the feasibility of GSK Biologicals' GSK2197870A vaccine co-administered with Wyeth-Lederle's Prevenar™ when given in healthy infants as a three-dose primary vaccination course at 2, 3 and 4 months of age followed by a booster dose of GSK Biologicals' Menitorix™ at 12 months of age.

DETAILED DESCRIPTION:
This protocol posting has been updated following Protocol amendment 1, 11-February-2010; The Study design section is impacted by this amendment.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry:

* A male or female infant between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Born after 36 to 42 weeks of gestation.
* Subjects who the investigator believes that their parents/ guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any apply, the subject must not be included in the study:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone, or equivalent, >= 0.5 mg/kg/day. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product .
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, poliomyelitis, Hib, pneumococcal and/or group C meningococcal vaccination or disease.
* History of seizures or progressive neurological disease (one episode of febrile convulsion does not constitute an exclusion criterion).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.

The following condition is temporary or self limiting and a subject may be vaccinated once the condition has resolved and no other exclusion criteria are met:

• Current febrile illness or axillary temperature ≥37.5ºC or other moderate to severe illness within 24 hours of study vaccine administration

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2009-06-24; Primary Completion 2010-03-31 (Actual); Study Completion 2010-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United Kingdom (5):
  - GSK Investigational Site, Ely, Cambridgeshire
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Oxford, Oxfordshire
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Khatami A, Snape MD, Ohene-Kena B, Young K, Oeser C, Michaelis LJ, Macleod E, Smee H, Van Der Meeren O, Leyssen M, Caubet M, Yu LM, Heath PT, Faust SN, Finn A, Pollard AJ. Phase II study of a three-dose primary vaccination course of DTPa-IPV/Hib-MenC-TT followed by a 12-month Hib-MenC-TT booster in healthy infants. Pediatr Infect Dis J. 2013 Jun;32(6):675-81. doi: 10.1097/INF.0b013e31828672a7. PMID 23348809
- [Background] Khatami A et al. Phase II study of a three-dose primary vaccination course of DTPa-IPV/Hib-MenC-TT followed by a 12-month Hib-MenC-TT booster in healthy infants. Abstract presented at the 7th World Congress World Society for Pediatric Infectious Diseases (WSPID). Melbourne, Australia, 16-19 November 2011.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111709 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111709 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111709 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111709 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111709 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111709 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111709 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 284 subjects were enrolled in the study.
Groups:
- GSK2197870A Group: Subjects aged between and including 6 and 12 weeks of age at the time of first vaccination received 3 doses of GSK2197870A vaccine at Months 0, 1 and 2, 2 doses of Prevenar vaccine at Months 0 and 2 and a booster dose of Menitorix vaccine at Month 10. All vaccines were administered intramuscularly. GSK2197870A and Menitorix vaccines were administered in the right upper anterolateral thigh and Prevenar vaccine in the left upper anterolateral thigh.
- Pediacel Group: Subjects aged between and including 6 and 12 weeks of age at the time of first vaccination received 3 doses of Pediacel vaccine at Months 0, 1 and 2, 2 doses of Prevenar vaccine at Months 0 and 2, 2 doses of Menjugate vaccine at Months 1 and 2 and a booster dose of Menitorix at Month 10. All vaccines were administered intramuscularly. Pediacel and Menitorix vaccines were administered in the right upper anterolateral thigh and Prevenar vaccine in the left upper anterolateral thigh and Menjugate vaccine in the left lower anterolateral thigh.
Period: Prior to Booster
Arm/Group | GSK2197870A Group | Pediacel Group
Started | 142 | 142
Completed | 140 | 139
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Period: After Booster
Arm/Group | GSK2197870A Group | Pediacel Group
Started | 139 | 135
Completed | 139 | 135
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2197870A Group | Pediacel Group | Total
Number analyzed (Participants) | 142 | 142 | 284
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Primary vaccination epoch Population: Baseline characteristics for primary vaccine population.
  weeks | 8.2 (0.69) | 8.1 (0.74) | 8.15 (0.49)
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Booster vaccination epoch Population: Baseline characteristics for booster vaccine population.
  weeks
    number analyzed (Participants) | 139 | 135 | 274
    (all) | 11.8 (0.39) | 11.9 (0.36) | 11.85 (0.38)
Sex: Female, Male [Count of Participants; unit: Participants] — Primary vaccination epoch Population: Baseline characteristics for primary vaccine population.
  Participants
    Female | 59 | 78 | 137
    Male | 83 | 64 | 147
Sex: Female, Male [Count of Participants; unit: Participants] — Booster vaccination epoch Population: Baseline characteristics for booster vaccine population.
  Participants
    number analyzed (Participants) | 139 | 135 | 274
    Female | 59 | 75 | 134
    Male | 80 | 60 | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Primary vaccination epoch Population: Baseline characteristics for primary vaccine population,
  Participants
    African Heritage/African American | 2 | 3 | 5
    Asian - Central/South Asian Heritage | 3 | 3 | 6
    Asian - East Asian Heritage | 2 | 1 | 3
    Asian - South East Asian Heritage | 1 | 1 | 2
    White - Caucasian/European Heritage | 121 | 130 | 251
    Other | 13 | 4 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Booster vaccination epoch Population: Baseline characteristics for booster vaccine population.
  Participants
    African Heritage/African American: number analyzed (Participants) | 139 | 135 | 274
    African Heritage/African American | 2 | 2 | 4
    American Indian or Alaskan Native: number analyzed (Participants) | 139 | 135 | 274
    American Indian or Alaskan Native | 0 | 0 | 0
    Asian - Central/South Asian Heritage: number analyzed (Participants) | 139 | 135 | 274
    Asian - Central/South Asian Heritage | 3 | 3 | 6
    Asian - East Asian Heritage: number analyzed (Participants) | 139 | 135 | 274
    Asian - East Asian Heritage | 1 | 1 | 2
    Asian - Japanese Heritage: number analyzed (Participants) | 139 | 135 | 274
    Asian - Japanese Heritage | 0 | 0 | 0
    Asian - South East Asian Heritage: number analyzed (Participants) | 139 | 135 | 274
    Asian - South East Asian Heritage | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 139 | 135 | 274
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    White - Arabic/North African Heritage: number analyzed (Participants) | 139 | 135 | 274
    White - Arabic/North African Heritage | 0 | 0 | 0
    White - Caucasian/European Heritage: number analyzed (Participants) | 139 | 135 | 274
    White - Caucasian/European Heritage | 119 | 124 | 243
    Other: number analyzed (Participants) | 139 | 135 | 274
    Other | 13 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects for Anti-polyribosylribitol Phosphate (Anti-PRP).
Description: A seroprotected subject was defined as a vaccinated subject who had anti-PRP antibody concentrations ≥ 0.15 micrograms per milliliter (µg/mL).
Time Frame: At Month 3
Population: The analysis was performed on the Primary According-To-Protocol cohort for immunogenicity, which included all evaluable subjects, for whom assay results were available for antibodies against at least one study vaccine antigen component after at least one vaccination during the primary vaccination course.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 108 | 119
Participants | 108 | 111

2. Primary Outcome: Number of Seropositive Subjects Against Neisseria Meningitidis Using Baby Rabbit Complement (rSBA-MenC)
Description: A seropositive subject was defined as a vaccinated subject who had rSBA-MenC ≥ 1:8.
Time Frame: At Month 2 and Month 3.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 109 | 113
Participants
  rSBA-MenC at Month 2 [N=109;111] | 104 | 109
  rSBA-MenC at Month 3 [N=105;113] | 101 | 113

3. Secondary Outcome: Number of Subjects With Anti-PRP Concentrations Antibody Above the Cut-off.
Description: The reference cut-off was ≥ 1.0 micrograms per milliliter (µg/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 108 | 119
Subjects | 96 | 98

4. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC ) Antibody Concentrations Above the Cut-offs.
Description: The reference cut-offs were ≥ 0.3 µg/mL and ≥ 2 µg/mL.
Time Frame: At Month 2 and Month 3.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 113 | 115
Subjects
  Anti-PSC ≥ 0.3 µg/mL at Month 2 [N=113;115] | 113 | 115
  Anti-PSC ≥ 0.3 µg/mL at Month 3 [N=108;114] | 108 | 114
  Anti-PSC ≥ 2.0 µg/mL at Month 2 [N=113;115] | 113 | 113
  Anti-PSC ≥ 2.0 µg/mL at Month 3 [N=108;114] | 107 | 114

5. Secondary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies.
Description: A seroprotected subject was defined as a vaccinated subject who had anti-D and anti-T antibody concentrations ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 3.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 108 | 119
Subjects
  Anti-T | 108 | 119
  Anti-D | 108 | 119

6. Secondary Outcome: Number of Seropositive Subjects Against Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN).
Description: A seropositive subject was defined as a vaccinated subject who had anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 enzyme-linked immunosorbent assay (ELISA) units per milliliters (EL.U/mL).
Time Frame: At Month 3.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 108 | 120
Subjects
  Anti-PT [N=107;117] | 107 | 117
  Anti-FHA [N=106;119] | 106 | 119
  Anti-PRN [N=108;120] | 108 | 119

7. Secondary Outcome: Number of Seroprotected Subjects for Anti-poliovirus (Anti-polio) Types 1, 2 and 3.
Description: A seroprotected subject was defined as a vaccinated subject who had anti-polio 1, 2 and 3 antibody concentrations ≥ 1:8.
Time Frame: At Month 3.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 89 | 94
Subjects
  Anti-polio 1 | 89 | 93
  Anti-polio 2 | 88 | 92
  Anti-polio 3 | 89 | 94

8. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal (Anti-PNE) Serotypes.
Description: A seropositive subject was defined as a vaccinated subject who had anti- pneumococcal antibody concentrations ≥ 0.2 micrograms per milliliter (µg/mL). The anti-PNE serotypes assessed were 4, 6B, 9V, 14, 18C, 19F and 23F.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 108 | 112
Subjects
  Anti- PNE 4 [N=47;52] | 47 | 52
  Anti- PNE 6B [N=46;52] | 14 | 13
  Anti- PNE 9V [N=47;51] | 46 | 49
  Anti- PNE 14 [N=47;52] | 47 | 50
  Anti- PNE 18C [N=46;52] | 45 | 51
  Anti- PNE 19F [N=47;52] | 46 | 52
  Anti- PNE 23F [N=47;52] | 37 | 49

9. Secondary Outcome: Concentrations for Anti-PRP.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection reference cut-off value was ≥ 0.15 µg/mL.
Time Frame: At Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 108 | 119
µg/mL | 4.347 [3.507 to 5.389] | 4.347 [3.507 to 5.389]

10. Secondary Outcome: Titers for rSBA-MenC.
Description: Titers were expressed as geometric mean titers (GMCs). The seropositivity reference cut-off value was ≥ 1:8.
Time Frame: At Month 2 and Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 109 | 113
titers
  rSBA-MenC at Month 2 [N=109;111] | 339.4 [254.5 to 452.7] | 257.0 [204.5 to 323.0]
  rSBA-MenC at Month 3 [N=105;113] | 393.2 [292.5 to 528.7] | 3110.5 [2612.0 to 3704.2]

11. Secondary Outcome: Concentrations for Anti-PSC.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection reference cut-off value was ≥ 0.3 µg/mL.
Time Frame: At Month 2 and Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 113 | 115
µg/mL
  Anti-PSC at Month 2 [N=113;115] | 18.20 [15.91 to 20.82] | 10.77 [9.61 to 12.08]
  Anti-PSC at Month 3 [N=108;114] | 15.10 [13.00 to 17.55] | 17.29 [15.53 to 19.25]

12. Secondary Outcome: Concentrations for Anti-T and Anti-D.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection reference cut-off value was ≥ 0.1 IU/mL.
Time Frame: At Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 108 | 119
IU/mL
  Anti-T | 2.694 [2.394 to 3.032] | 1.034 [0.895 to 1.195]
  Anti-D | 1.767 [1.548 to 2.019] | 1.817 [1.589 to 2.078]

13. Secondary Outcome: Concentrations for Anti-PT, Anti-FHA and Anti-PRN.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seropositivity reference cut-off value was ≥ 5 EL.U/mL.
Time Frame: At Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 108 | 120
EL.U/mL
  Anti-PT [N=107;117] | 45.4 [40.0 to 51.4] | 45.1 [39.8 to 51.2]
  Anti-FHA [N=106;119] | 234.4 [203.7 to 269.6] | 204.9 [178.2 to 235.6]
  Anti-PRN [N=108;120] | 121.6 [103.6 to 142.7] | 49.9 [41.4 to 60.1]

14. Secondary Outcome: Titers for Anti-polio 1, 2 and 3.
Description: Titers were expressed as geometric mean titers (GMTs). The seropositivity reference cut-off value was ≥ 1:8.
Time Frame: At Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 89 | 94
titers
  Anti-polio 1 | 169.4 [127.0 to 226.0] | 89.3 [71.1 to 112.2]
  Anti-polio 2 | 90.2 [68.5 to 118.7] | 77.7 [59.7 to 101.1]
  Anti-polio 3 | 367.9 [288.1 to 469.9] | 250.5 [195.9 to 320.2]

15. Secondary Outcome: Concentrations for Anti-PNE Serotypes.
Description: Concentrations were expressed as geometric mean concentreations (GMCs). The seropositivity reference cut-off value was ≥ 0.2 µg/mL.
Time Frame: At Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 89 | 94
µg/mL
  Anti- PNE 4 [N=47;52] | 2.56 [2.13 to 3.07] | 2.18 [1.87 to 2.53]
  Anti- PNE 6B [N=46;52] | 0.12 [0.08 to 0.17] | 0.12 [0.08 to 0.16]
  Anti- PNE 9V [N=47;51] | 2.56 [1.92 to 3.43] | 1.85 [1.43 to 2.39]
  Anti- PNE 14 [N=47;52] | 3.78 [2.70 to 5.28] | 2.71 [2.00 to 3.67]
  Anti- PNE 18C [N=46;52] | 2.26 [1.59 to 3.20] | 2.74 [2.12 to 3.56]
  Anti- PNE 19F [N=47;52] | 3.00 [2.21 to 4.06] | 3.15 [2.51 to 3.95]
  Anti- PNE 23F [N=47;52] | 0.58 [0.40 to 0.82] | 0.89 [0.69 to 1.14]

16. Secondary Outcome: Number of Seroprotected Subjects for Anti-PRP.
Description: as for outcome 1
Time Frame: At Month 10 and Month 11.
Population: The analysis was performed on the Booster According-To-Protocol cohort for immunogenicity, which included all evaluable subjects, for whom assay results were available for antibodies against at least one study vaccine antigen for the blood sample taken 30 days after the administration of the booster vaccination course.
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 98 | 112
Subjects
  Anti-PRP at Month 10 [N=89;98] | 76 | 81
  Anti-PRP at Month 11 [N=98;112] | 98 | 112

17. Secondary Outcome: Number of Seropositive Subjects Against rSBA-MenC.
Description: A seropositive subject was defined as a vaccinated subject who had rSBA-MenC ≥ 1:8.
Time Frame: At Month 10 and Month 11.
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 94 | 109
Subjects
  rSBA-MenC at Month 10 [N=87;93] | 70 | 78
  rSBA-MenC at Month 11 [N=94;109] | 93 | 109

18. Secondary Outcome: Number of Subjects With Anti-PSC Antibody Concentrations Above the Cut-offs.
Description: The reference cut-offs were ≥ 0.3 µg/mL and ≥ 2 µg/mL.
Time Frame: At Month 10 and Month 11.
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 100 | 111
Subjects
  Anti-PSC ≥ 0.3 µg/mL at Month 10 [N=86;97] | 81 | 89
  Anti-PSC ≥ 0.3 µg/mL at Month 11 [N=100;111] | 100 | 111
  Anti-PSC ≥ 2.0 µg/mL at Month 10 [N=86;97] | 22 | 14
  Anti-PSC ≥ 2.0 µg/mL at Month 11 [N=100;111] | 92 | 80

19. Secondary Outcome: Number of Seroprotive Subjects for Anti-D and Anti-T Antibodies.
Description: A seropositive subject was defined as a vaccinated subject who had anti-D (ELISA) and anti-T antibody concentrations ≥ 0.1 IU/mL. Seropositivity for anti-D was also defined with the ≥ 0.016 IU/mL cut-off (Neutralisation assay).
Time Frame: At Month 10.
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 89 | 98
Subjects
  Anti-T ≥ 0.1 IU/mL [N=89;98] | 86 | 87
  Anti-D ≥ 0.1 IU/mL [N=89;98] | 72 | 94
  Anti-D ≥ 0.016 IU/mL [N=16;3] | 11 | 3

20. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN.
Description: as for outcome 6
Time Frame: At Month 10.
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 89 | 100
Subjects
  Anti-PT [N=89;100] | 60 | 88
  Anti-FHA [N=89;99] | 89 | 98
  Anti-PRN [N=89;100] | 75 | 72

21. Secondary Outcome: Number of Seroprotected Subjects for Anti-anti-polio Types 1, 2 and 3.
Description: A seroprotected subject was defined as a vaccinated subject who had anti-polio 1, 2 and 3 antibody concentrations ≥ 1:8.
Time Frame: At Month 10.
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 78 | 86
Subjects
  Anti-polio 1 [N=78;86] | 68 | 62
  Anti-polio 2 [N=78;85] | 63 | 69
  Anti-polio 3 [N=78;86] | 74 | 76

22. Secondary Outcome: Concentrations for Anti-PRP.
Description: as for outcome 9
Time Frame: At Month 10 and Month 11.
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: µg /mL
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 98 | 112
µg /mL
  Anti-PRP at Month 10 [N=89;98] | 0.423 [0.339 to 0.528] | 0.574 [0.436 to 0.756]
  Anti-PRP at Month 11 [N=98;112] | 66.697 [53.271 to 83.507] | 26.899 [20.931 to 34.569]

23. Secondary Outcome: Titers for rSBA-MenC.
Description: Titers were expressed as geometric mean titers (GMCs). The seropositivity reference cut-off value was ≥ 1:8.
Time Frame: At Month 10 and Month 11.
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 93 | 109
titers
  rSBA-MenC at Month 10 [N=87;94] | 62.1 [43.3 to 89.1] | 67.1 [48.5 to 92.7]
  rSBA-MenC at Month 11 [N=93;109] | 3062.9 [2421.2 to 3874.6] | 954.0 [761.3 to 1195.5]

24. Secondary Outcome: Concentrations for Anti-PSC.
Description: as for outcome 11
Time Frame: At Month 10 and Month 11.
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: µg /mL
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 100 | 111
µg /mL
  Anti-PSC at Month 10 [N=86;97] | 0.94 [0.76 to 1.15] | 0.87 [0.74 to 1.04]
  Anti-PSC at Month 11 [N=100;111] | 6.15 [5.24 to 7.22] | 2.88 [2.49 to 3.32]

25. Secondary Outcome: Concentrations for Anti-T and Anti-D.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection reference cut-off value was ≥ 0.1 IU/mL. Seropositivity for anti-D was also defined with the ≥ 0.016 IU/mL cut-off (Neutralisation assay).
Time Frame: At Month 10.
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 89 | 98
IU/mL
  Anti-T ≥ 0.1 IU/mL [N=89;98] | 0.428 [0.361 to 0.508] | 0.260 [0.217 to 0.311]
  Anti-D ≥ 0.1 IU/mL [N=89;98] | 0.249 [0.202 to 0.307] | 0.385 [0.330 to 0.448]
  Anti-D ≥ 0.016 IU/mL [N=16;3] | 0.015 [0.012 to 0.020] | 0.020 [0.008 to 0.052]

26. Secondary Outcome: Concentrations for Anti-PT, Anti-FHA and Anti-PRN.
Description: as for outcome 13
Time Frame: At Month 10.
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 89 | 100
EL.U/mL
  Anti-PT [N=89;100] | 7.3 [6.1 to 8.8] | 9.8 [8.5 to 11.4]
  Anti-FHA [N=89;99] | 35.3 [28.3 to 44.0] | 48.8 [40.4 to 58.9]
  Anti-PRN [N=89;100] | 15.0 [11.8 to 19.0] | 9.6 [7.7 to 11.9]

27. Secondary Outcome: Titers for Anti-polio 1, 2 and 3.
Description: Titers were expressed as geometric mean titers (GMTs). The seroprotection reference cut-off value was ≥ 1:8.
Time Frame: At Month 10.
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 78 | 89
titers
  Anti-polio 1 [N=78;86] | 36.3 [26.5 to 49.8] | 18.8 [14.4 to 24.7]
  Anti-polio 2 [N=78;85] | 28.5 [20.9 to 39.0] | 24.5 [18.8 to 32.0]
  Anti-polio 3 [N=78;86] | 70.1 [51.0 to 96.3] | 50.7 [37.0 to 69.4]

28. Secondary Outcome: Number of Subjects With a Booster Response to rSBA-MenC Antibodies.
Description: Booster response defined as: for initially seronegative subjects, antibody titre ≥ 1:32 at post-booster (Month 11); for initially seropositive subjects, antibody titres at post-booster ≥ 4 fold the pre-booster.
Time Frame: At Month 11
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 71 | 79
Subjects | 68 | 61

29. Secondary Outcome: Number of Subjects With a Booster Response to Anti-PRP Antibodies.
Description: Booster response defined as: for initially seronegative subjects, antibody concentration ≥ 0.6 µg/mL at post-booster (Month 11); for initially seropositive subjects, antibody concentrations at post-booster ≥ 4 fold the pre-booster.
Time Frame: At Month 11
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 75 | 87
Subjects | 75 | 85

30. Secondary Outcome: Number of Subjects With a Booster Response to Anti-PSC Antibodies.
Description: Booster response defined as: for initially seronegative subjects, antibody concentration ≥ 1.2 µg/mL at post-booster (Month 11); for initially seropositive subjects, antibody concentrations at post-booster ≥ 4 fold the pre-booster.
Time Frame: At Month 11
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 75 | 83
Subjects | 48 | 27

31. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7)
Population: The analysis was performed on the Primary Total Vaccinated cohort, which included all subjects with at least one study vaccine administration documented during the primary course.
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 142 | 141
Subjects
  Any pain | 57 | 57
  Any redness | 86 | 77
  Any swelling | 60 | 48

32. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms.
Description: as for outcome 31
Time Frame: During the 8-day (Days 0-7)
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all subjects vaccinated with the booster dose.
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 136 | 134
Subjects
  Any pain | 24 | 11
  Any redness | 74 | 56
  Any swelling | 35 | 20

33. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms.
Description: Solicited general symptoms assessed were drowsiness, irritability, loss of appetite and fever [axillary temperature above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7)
Population: as for outcome 31
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 142 | 141
Subjects
  Any drowsiness | 103 | 103
  Any irritability | 122 | 117
  Any loss of appetite | 79 | 77
  Any fever | 59 | 49

34. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms.
Description: as for outcome 33
Time Frame: During the 8-day (Days 0-7)
Population: as for outcome 32
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 136 | 134
Subjects
  Any drowsiness | 43 | 40
  Any irritability | 75 | 66
  Any loss of appetite | 41 | 40
  Any fever | 18 | 20

35. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of an AE regardless of intensity grade or relationship to study vaccination.
Time Frame: Within the 31-day (Days 0-30) follow up period after vaccination.
Population: as for outcome 31
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 142 | 142
Subjects | 114 | 112

36. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: as for outcome 35
Time Frame: Within the 31-day (Days 0-30) follow up period after vaccination.
Population: as for outcome 32
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 139 | 135
Subjects | 75 | 66

37. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization or results in disability/incapacity of a study subjects. Any SAE = any SAE regardless of assessment of relationship to study vaccination.
Time Frame: During the entire study period (Month 0 to Month 11)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | GSK2197870A Group | Pediacel Group
Number analyzed (Participants) | 142 | 142
Subjects | 9 | 6

ADVERSE EVENTS:
Time Frame: Solicited symptoms: 8-day follow-up period after vaccination; unsolicited AEs: 31-day follow-up period after vaccination; SAEs: during the entire study period (Months 0-11).
Arm/Group | GSK2197870A Group | Pediacel Group
Serious Adverse Events (participants affected / at risk) | 9/142 | 6/142
Other Adverse Events (participants affected / at risk) | 141/142 | 141/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2197870A Group (N=142) | Pediacel Group (N=142)
Bronchiolitis (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Developmental delay (General disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lymph node abscess (Blood and lymphatic system disorders) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4.9% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2197870A Group (N=142) | Pediacel Group (N=142)
Rhinitis (Infections and infestations) | 42 | 35 — Symptom reported during the primary phase.
Teething (Gastrointestinal disorders) | 31 | 29 — Symptom reported during the primary phase.
Diarrhoea (Gastrointestinal disorders) | 19 | 18 — Symptom reported during the primary phase.
Vomiting (Gastrointestinal disorders) | 21 | 14 — Symptom reported during the primary phase.
Nasopharyngitis (Infections and infestations) | 13 | 18 — Symptom reported during the primary phase.
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 15 — Symptom reported during the primary phase.
Eczema (Skin and subcutaneous tissue disorders) | 7 | 14 — Symptom reported during the primary phase.
Upper respiratory tract infection (Infections and infestations) | 6 | 8 — Symptom reported during the primary phase.
Teething (Gastrointestinal disorders) | 28/139 | 23 — Symptom reported during the booster phase.
Rash (General disorders) | 7/139 | 9 — Symptom reported during the booster phase.
Nasopharyngitis (Infections and infestations) | 11/139 | 2 — Symptom reported during the booster phase.
Diarrhoea (Gastrointestinal disorders) | 5/139 | 7 — Symptom reported during the booster phase.
Upper respiratory tract infection (Infections and infestations) | 5/139 | 7 — Symptom reported during the booster phase.
Pain (General disorders) | 57 | 57/141 — Symptom reported during the primary phase.
Redness (General disorders) | 86 | 77/141 — Symptom reported during the primary phase.
Swelling (General disorders) | 60 | 48/141 — Symptom reported during the primary phase.
Pain (General disorders) | 24 | 11/134 — Symptom reported during the booster phase.
Redness (General disorders) | 76 | 56/134 — Symptom reported during the booster phase.
Swelling (General disorders) | 35 | 20/134 — Symptom reported during the booster phase.
Drowsiness (General disorders) | 103 | 103/141 — Symptom reported during the primary phase.
Irritability (General disorders) | 122 | 117/141 — Symptom reported during the primary phase.
Loss of appetite (General disorders) | 79 | 77/141 — Symptom reported during the primary phase.
Fever (General disorders) | 59 | 49/141 — Symptom reported during the primary phase.
Drowsiness (General disorders) | 43/136 | 40/134 — Symptom reported during the booster phase.
Irritability (General disorders) | 75/136 | 66/134 — Symptom reported during the booster phase.
Loss of appetite (General disorders) | 41/136 | 40/134 — Symptom reported during the booster phase.
Fever (General disorders) | 18/136 | 20/134 — Symptom reported during the booster phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.